CLINICAL TRIAL: NCT02191930
Title: Brentuximab Vedotin or B-CAP in the Treatment of Older Patients With Newly Diagnosed Classical Hodgkin Lymphoma - a GHSG-NLG Intergroup Phase II Trial -
Brief Title: Brentuximab Vedotin or B-CAP in the Treatment of Older Patients With Newly Diagnosed Classical Hodgkin Lymphoma
Acronym: BVB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Prof., University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1707
Record Dates: First submitted 2014-07-11; First posted 2014-07-16 (Estimated); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Cyclophosphamide; Doxorubicin

ARMS (2):
- B-CAP (Experimental): Patients with ECOG of 2 or less (3 or less if caused by HL) and CIRS-G score of 6 or less (overall) and 3 or less per organ system receive 6 cycles of B-CAP (Brentuximab vedotin, cyclophosphamide, doxorubicine, predniso(lo)ne). Cycle length is 21 days
  Interventions: Drug: B-CAP
- Brentoximab Vedotin only (Experimental): Patients with CIRS-G score of 7 ore more receive Brentuximab Vedotin as single agent therapy for up to 16 cycles. Cycle length is 21 days
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: B-CAP
  Other Names: Brentuximab Vedotin; Cyclophosphamide; Doxorubicine; Predniso(lo)ne
  Arms: B-CAP
Drug: Brentuximab Vedotin
  Arms: Brentoximab Vedotin only

SUMMARY:
The purpose of this trial is to determine

1. Objective response rate (ORR), defined as the proportion of patients having CR, CRr or PR in the centrally reviewed restaging after six cycles of chemotherapy
2. Progression-free survival (PFS) 3 years after registration

ELIGIBILITY:
Inclusion Criteria (B-CAP):

* classical Hodgkin Lymphoma
* Age 60 years or older
* ECOG performance status ≤ 2 or ≤ 3 if due to HL
* CIRS-G score of ≤ 6 and ≤ 3 per organ system (except score 4 for eye, ear, nose and throat)
* Advanced stages: Stage IIB with large mediastinal mass and/or extranodal lesions, stage III or IV disease
* written informed consent

Exclusion Criteria (B-CAP):

* Composite lymphoma or nodular lymphocyte- predominant Hodgkin lymphoma (NLPHL)
* Prior chemotherapy or radiation for HL except prephase
* Peripheral neuropathy greater than CTC Grade 1

Inclusion Criteria (BV only):

* classical Hodgkin Lymphoma
* Age 60 years or older
* stage IA to IVB
* CIRS-G score of ≥ 7 or 4 in one organ system (except score 4 for eye, ear, nose and throat)
* Patients not eligible to curative poly-chemotherapy at the investigators judgment
* written informed consent

Exclusion Criteria (BV only):

* Composite lymphoma or nodular lymphocyte- predominant Hodgkin lymphoma (NLPHL)
* Prior chemotherapy or radiation for HL except prephase as outlined in the protocol
* Peripheral neuropathy greater than CTC Grade 1

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate | after 6 cycles of therapy (at least 18 weeks after start of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof., Principal Investigator — University Hospital of Cologne
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- See also: Homepage GHSG — http://www.ghsg.org